CLINICAL TRIAL: NCT05040256
Title: Neurologic and Immunologic Characteristics of CTLA-4 and LRBA Hereditary Deficiency
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0290
Record Dates: First submitted 2021-05-11; First posted 2021-09-10 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: CTLA4 Haploinsufficiency
Keywords: LRBA deficiency; Primary immunodeficiency; Neuroinflammation; Genetic diseases; Autoimmune diseases
MeSH Terms: conditions — Diabetes Mellitus, Insulin-Dependent, 12; Primary Immunodeficiency Diseases; Neuroinflammatory Diseases; Genetic Diseases, Inborn; Autoimmune Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
CTLA4 and LRBA deficiencies are rare genetic disorders, recently described, and associated with multiple clinical features. It ranges from recurrent infections, auto-immunity, and organ infiltration with lymphocytes. Neurologic syndroms are described in up to 30% of patients, yet they are poorly defined to date. Early recognition of a specific pattern can be important, given that there is a targeted therapy in this situation.

ELIGIBILITY:
Inclusion criteria:

- Patients diagnosed with CTLA4 or LRBA mutation

Exclusion criteria:

- Age < 12 years

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients listed with CTLA4 or LRBA deficiency in the register of the national reference center for primary immunodeficiencies.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Number of Neurologic impairment | 1 day
  Neurologic signs and symptoms (headaches, seizures…), cerebral MRI features, lumbar puncture, histopathology

SECONDARY OUTCOMES:
Presence of reccurent infections | 1 day
  Presence of reccurent infections and type, granulomatous disease, cancer predisposition, immunologic biological tests, type of treatments and effectiveness

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Ayrignac, MD, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC

REFERENCES:
- [Result] Schindler MK, Pittaluga S, Enose-Akahata Y, Su HC, Rao VK, Rump A, Jacobson S, Cortese I, Reich DS, Uzel G. Haploinsufficiency of immune checkpoint receptor CTLA4 induces a distinct neuroinflammatory disorder. J Clin Invest. 2020 Oct 1;130(10):5551-5561. doi: 10.1172/JCI135947. PMID 32955488
- [Result] Ayrignac X, Goulabchand R, Jeziorski E, Rullier P, Carra-Dalliere C, Lozano C, Portales P, Vincent T, Viallard JF, Menjot de Champfleur N, Rieux-Laucat F, Besnard C, Koenig M, Guissart C, Labauge P, Guilpain P. Two neurologic facets of CTLA4-related haploinsufficiency. Neurol Neuroimmunol Neuroinflamm. 2020 Jun 4;7(4):e751. doi: 10.1212/NXI.0000000000000751. Print 2020 Jul. PMID 32499327
- [Result] Schubert D, Bode C, Kenefeck R, Hou TZ, Wing JB, Kennedy A, Bulashevska A, Petersen BS, Schaffer AA, Gruning BA, Unger S, Frede N, Baumann U, Witte T, Schmidt RE, Dueckers G, Niehues T, Seneviratne S, Kanariou M, Speckmann C, Ehl S, Rensing-Ehl A, Warnatz K, Rakhmanov M, Thimme R, Hasselblatt P, Emmerich F, Cathomen T, Backofen R, Fisch P, Seidl M, May A, Schmitt-Graeff A, Ikemizu S, Salzer U, Franke A, Sakaguchi S, Walker LSK, Sansom DM, Grimbacher B. Autosomal dominant immune dysregulation syndrome in humans with CTLA4 mutations. Nat Med. 2014 Dec;20(12):1410-1416. doi: 10.1038/nm.3746. Epub 2014 Oct 20. PMID 25329329